CLINICAL TRIAL: NCT00530153
Title: School Intervention Study of Nutrition, Wellbeing and Dental Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: University of Oulu, Department of dental health (Other); Sitra, the Finnish Innovation Fund (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KTL 369-3
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Eating; Oral Health
Keywords: Eating; Food Habits; Adolescent; Dental Research
MeSH Terms: conditions — Feeding Behavior | interventions — Nutrition Assessment; Xylitol

INTERVENTIONS:
Behavioral: dietary counseling — Various activities and materials for teachers, students, parents and school catering personnel aiming at increasing their awareness and knowledge of good nutrition.
Dietary Supplement: xylitol — Delivery of xylitol lozenges (about 1 g xylitol/student/school day) and guidance on tooth brushing.

SUMMARY:
The purpose of this study is to evaluate the effects of an intervention programme on dietary intake and dental health of 8th grade students.

ELIGIBILITY:
Inclusion Criteria:

* 7th grade students from the participating schools, written informed consent both from the student and the parent

Ages: 13 Years to 14 Years | Sex: All
Age Groups: Child
Enrollment: 769 (Actual)
Dates: Start 2007-04; Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Dietary intake (eg. sugar, fibre). The presence of active initial caries lesions.

SECONDARY OUTCOMES:
Nutritional quality of school meals and snacks. Laser fluorescence values of the occlusal surfaces of permanent molar and premolar teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Pietinen, Ph. D, Principal Investigator — National Public Health Institute
Locations (1):
- National Public Health Institute, Helsinki, Finland